CLINICAL TRIAL: NCT01599494
Title: A Multi-center, Open-label, Randomized Trial in India to Investigate the Efficacy and Safety of a Single Injection of MK-8962 (Corifollitropin Alfa) to Induce Multifollicular Development for Controlled Ovarian Stimulation Using Daily Recombinant FSH as a Reference (Phase III, Protocol No. MK-8962-029-00 [Also Known as SCH900962, P07056])
Brief Title: An Efficacy and Safety Study of Corifollitropin Alfa (MK-8962) in Contrast to Recombinant FSH for Use in Controlled Ovarian Stimulation of Indian Women (P07056, Also Known as MK-8962-029)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P07056; MK-8962-029 (Other: Merck)
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta; ganirelix; Chorionic Gonadotropin; Progesterone; Crinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-Dose MK-8962 + recFSH (Experimental)
  Interventions: Drug: MK-8962; Drug: recFSH; Drug: Ganirelix; Drug: human Chorionic Gonadotropin (hCG); Drug: Progesterone
- Reference Group recFSH only (Active Comparator)
  Interventions: Drug: recFSH; Drug: Ganirelix; Drug: human Chorionic Gonadotropin (hCG); Drug: Progesterone

INTERVENTIONS:
Drug: MK-8962 — MK-8962 is supplied in a ready-to-use prefilled syringe containing
  100 microgram (μg) or 150 μg corifollitropin alfa per 0.5 mL. Participants are randomized to receive a single subcutaneous (SC) injection of MK-8962 in the abdominal wall on Cycle Day 2 or Cycle Day 3. Dose of administered MK-8962 is weight-based. Participants who weigh 60 kilograms (kg) or less will be given 100 μg MK-8962 and those who weigh more than 60 kg will be given 150 μg MK-8962.
  Other Names: Corifollitropin alfa
  Arms: Single-Dose MK-8962 + recFSH
Drug: recFSH — Recombinant Follicle Stimulating Hormone (recFSH) will be supplied as a ready-to-use solution in a 600 IU cartridge for SC injection via the recFSH Pen. Starting on Day 2 or 3 of the menstrual cycle (Stimulation Day 1), recFSH will be administered daily, each morning, via injections in the abdominal wall. A starting dose of between 150 - 300 IU will be administered and is fixed for the first week of stimulation. After 6 days, and based on each participant's individual response, the Investigator may decide to reduce the fixed dose for the remainder of the study. The maximum duration of stimulation is 19 days; recFSH will not be administered on the Day of hCG Administration.
  Other Names: follitropin beta
Drug: Ganirelix — 0.25 mg/day SC injection in the upper leg, administered on Stimulation Day 5 up to and including Day of hCG Administration
  Other Names: Ganirelix acetate or Ganirelix diacetate
Drug: human Chorionic Gonadotropin (hCG) — Single dose of 10,000 or 5,000 IU hCG, administered via SC injection on Day of hCG Administration.
  Other Names: human Chorionic Gonadotrophin
Drug: Progesterone — Crinone 8% (90 mg) gel administered intravaginally via a single-use, one piece polyethylene vaginal applicator once-daily on Day of Oocyte Pick-up or 1 day later and continued for at least 6 weeks or either up to menses or up to a negative pregnancy test performed at least 18 days after Day of Oocyte Pick-up.
  Other Names: Crinone®

SUMMARY:
This study, conducted in India, will be recruiting women participants who are between the ages of 18 and 42, and who have an indication for controlled ovarian stimulation (COS), but have not yet undergone in-vitro fertilization and/or intracytoplasmic sperm injection (IVF/ICSI). The study is designed to compare the difference in oocyte (immature egg cell) production after administration of the investigative drug, MK-8962 (corifollitropin alfa) + recombinant follicle stimulating hormone (recFSH), in contrast to use of only the reference drug, recFSH.

ELIGIBILITY:
Inclusion Criteria:

Please Note: In this trial an Indian female participant is defined as a woman 1) with native Indian parents, and 2) who is also in possession of an Indian identification card.

* Indian woman with an indication for COS and IVF/ICSI, but has not yet undergone IVF/ICSI.
* Body mass index (BMI) of 18.0 to 32.0 kg/m2
* Regular spontaneous menstrual cycle (ie, a menstrual schedule that consistently occurs within a range of 24 to 35 days)
* Access to available ejaculatory sperm. Use of donated and/or cryopreserved sperm is allowed, however sperm obtained via surgical sperm retrieval is not allowed.
* Results documented as 'within normal limits' from clinical laboratory tests (ie, complete blood count [CBC], blood chemistries, and urinalysis).
* Normal cervical smear result obtained within 12 months prior to study enrollment, otherwise test will be performed during screening.
* Able to adhere to dose and study visit schedules

Exclusion Criteria:

- Has a recent (ie, within 3 years prior to enrollment in study) history of/or

any active endocrine abnormality, treated or untreated.

* Contraindicated use of gonadotropins
* History of ovarian hyper-responsiveness
* History of/or current polycystic ovary syndrome (PCOS)
* Has less than 2 ovaries or has any other ovarian abnormality, including endometrioma (greater than 10 mm in size), and/or has unilateral or bilateral hydrosalpinx and/or intrauterine fibroids (5 cm in size or greater), confirmed by an ultrasound scan.
* Has any clinically relevant pathology that may impair embryo implantation or continuation of pregnancy.
* Experienced more than three unsuccessful COS cycles for IVF/ICSI since

the last established ongoing pregnancy, if applicable.

* History of non- or low ovarian response to FSH and/or Menopausal Gonadotropin (hMG) treatment.
* History of recurrent miscarriage (ie, 3 or more)
* Positive test results for Human Immunodeficiency Virus (HIV) or

Hepatitis B

* Recent history of/or current epilepsy, thrombophilia, diabetes, cardiovascular, gastro-intestinal, hepatic, renal or pulmonary or auto-immune disease, any of which required or requires treatment.
* Smokes or recently stopped smoking (ie, within 3 months of study enrollment)
* History of/or active alcohol and/or drug abuse (ie, within 12 months prior to study enrollment).
* Previous use of corifollitropin alfa
* Use of hormonal agents known to affect ovulation or any drug/agent considered to be teratogenic
* Use of any experimental drug within 3 months prior to study enrollment or participation in another clinical study, other than one that is survey-questionnaire based.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Number of Cumulus-Oocyte-Complexes Retrieved During Oocyte Pick-up | 34 to 36 hours after Day of Administration of Human Chorionic Gonadotropin (hCG)
  The criterion of hCG administration is defined as three or more follicles ≥17 mm, confirmed by ultrasound. Oocyte pick up occurs 34-36 hours after the Day of hCG Administration, based on confirmed ultrasound findings.

SECONDARY OUTCOMES:
Confirmation of Vital Pregnancy | Post treatment; at 35 days from Day of Embryo Transfer
  Per study protocol, vital pregnancy is defined as the presence of at least one fetus with heart activity at approximately 5 weeks (ie, ~ 35 days) after Day of Embryo Transfer in the COS treatment cycle.
Percentage of Participants with Moderate or Severe Ovarian Hyperstimulation Syndrome (OHSS) | From Baseline up to 10 weeks after Day of Embryo Transfer
  Per study protocol, OHSS is defined as more than 30 follicles ≥11 mm in size demonstrated by ultrasound.
Number of Participants with an Ongoing Pregnancy | Post treatment; at approximately 10 weeks from Day of Embryo Transfer
  Per study protocol, ongoing pregnancy is defined as confirmed pregnancy at 10 or more weeks ( ~ 70 days) after Day of Embryo Transfer, documented by a positive pregnancy test and ultrasound scan demonstrating at least one gestational sac with heart activity.